CLINICAL TRIAL: NCT05002049
Title: Science Engagement to Empower Disadvantaged adoleScents (SEEDS Project)
Acronym: SEEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: University of Exeter (Other); Harokopio University (Other); City of Rotterdam (Unknown); European Citizen Science Association (Unknown); Erasmus Medical Center (Other); Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SEEDS
Record Dates: First submitted 2021-07-15; First posted 2021-08-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy Lifestyle
Keywords: Healthy Lifestyle; Science Interest; Adolescents; Deprived; Citizen Science

STUDY DESIGN:
Intervention Model Description: High schools located in deprived areas will be randomized to the intervention group (IG) which will receive the whole citizen science intervention of the SEEDS project, or the controls group (CG) which will not receive any kind of intervention. As the high-schools will be the unit of randomization, this study is a cluster-randomized.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citizen Science Behavioral Intervention (Experimental): The intervention group (IG) participants will receive the whole citizen science intervention of the SEEDS project, and participants will be assessed at baseline and end-of-study.
  Interventions: Behavioral: Intervention Group
- Control Group (No intervention) (No Intervention): The controls group (CG) participants will not receive any kind of intervention, and participants will only be assessed at baseline and end-of-study.

INTERVENTIONS:
Behavioral: Intervention Group — Teenagers with leadership skills from intervention schools (called ambassadors) and stakeholders will participate in focus groups to gain insights on the barriers and facilitators for healthy lifestyles of teenagers, and how science could help address these. Building on the information of the focus groups, ambassadors, stakeholders and other peers will participate in a collaborative competition event where the SEEDS intervention(s) will be designed. The intervention(s) will be implemented at intervention high-schools during 6 months. Outcomes in health behaviours and science literacy will be assessed by validated questionnaires at the start and end of the project.
  Arms: Citizen Science Behavioral Intervention

SUMMARY:
SEEDS is a multicenter 24-month citizen science (CS) cluster randomized controlled study, with interventions conducted in four European countries acting as pilot sites: 1) Greece, 2) The Netherlands, 3) Spain and 4) The United Kingdom. This project will merge CS and traditional approaches and will target high schools located in deprived neighborhoods.

The methodology, that combines CS and traditional science, could build effective cooperation between science and society to empower adolescents from low-income environments to adopt healthy lifestyles to prevent obesity, increase their interest in science and improve their critical thinking.

DETAILED DESCRIPTION:
SEEDS is a multicenter 24-month citizen science (CS) cluster randomized controlled study, with interventions conducted in four European countries acting as pilot sites: 1) Greece, 2) The Netherlands, 3) Spain and 4) The United Kingdom. This project will merge CS and traditional approaches and will target high schools located in deprived neighborhoods.

The methodology, that combines CS and traditional science, could build effective cooperation between science and society to empower adolescents from low-income environments to adopt healthy lifestyles to prevent obesity, increase their interest in science and improve their critical thinking.

The aim is to engage teenagers on this citizen science project to collaborate in all phases of the study: problem definition, data collection, analyses and dissemination. This will empower them to change habits, thereby contributing to behavioural changes. This cluster-randomized control trial involves intervention and control high-schools from deprived areas in the Netherlands, England, Greece and Spain. Teenagers with leadership skills from intervention schools (called ambassadors) and stakeholders will participate in focus groups to gain insights on the barriers and facilitators for healthy lifestyles of teenagers, and how science could help address these. Building on the information of the focus groups, ambassadors, stakeholders and other peers will participate in a collaborative competition event where the SEEDS intervention(s) will be designed. The intervention(s) will be implemented at intervention high-schools. Outcomes in health behaviours and science literacy will be assessed by validated questionnaires at the start and end of the project.

ELIGIBILITY:
Inclusion Criteria per high schools:

* High schools located in deprived areas. Deprived areas will be selected according to what is considered an area with a low socioeconomic level according to each country.
* Informed consent must be signed by the responsible of each high-school.

Exclusion Criteria per high schools:

* The non-completion of one of the inclusion criteria.

Inclusion Criteria per participants:

* Adolescents aged 13- to 15-years at baseline who attended one of the participating high schools, previously randomized.
* Informed consent must be signed by their parents/legal guardians and by each adolescent.

Exclusion Criteria per participants:

* The non-completion of one of the inclusion criteria.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from Baseline to end-of-study (6-month)
  Change in physical activity assessed by validated questionnaire HBSC and Physical Activity Questionnaire for Children (PAQ-C).
  HBSC: days a week physically active for a total of at least 60 minutes, frequency of exercise in free time that participants get out of breath or sweat and means of transport to go to school.
  PAQ-C: 7-day recall questionnaire that assesses participation in different physical activities, as well as activity during Physical Education, lunch break, recess, after school, in the evenings and at weekends. Each of the 9 questionnaire items is scored between 1 (low) and 5 (high physical activity), and a mean score of all items constitutes the overall PAQ score.
Snacking choices | Change from Baseline to end-of-study (6-month)
  Change in healthy snacking choices (inside and outside school). This outcome will be assessed by validated questionnaires HBSC (times per week consume healthy and unhealthy snacking choices) and Beverage Frequency Questionnaire ( 7-day food record of beverages). Additionally, questions for assessing the frequency of consumption (times per week and time frame of the day) of each type of snack (chocolates, fruit and vegs, cakes or cookies and chocolates and sweets).
Sedentary time | Change from Baseline to end-of-study (6-month)
  Change in prolonged sedentary time. This outcome will be assessed by validated questionnaire HBSC (hours/day spend watching television/ playing computer games/ on computer for purposes other than playing).
Youth interest in life science | Change from Baseline to end-of-study (6-month)
  Changes in life science interest. This outcome will be measure by STEM interest survey.
Science capital perception and interest | Change from Baseline to end-of-study (6-month)
  Changes in science capital.This outcome will be measure by Science Capital Survey, developed by Archer et al. (2015): The selection of questions includes 4 components of the total Science Capital Survey: Future science job affinity (aspirations), utility of science qualifications, valuing science and scientists, and self-efficacy in science.
Youth interest in science technology engineering and math (STEM) career. | Change from Baseline to end-of-study (6-month)
  Changes in STEM career. This outcome will be measure by Attitude towards STEM questionnaire.

SECONDARY OUTCOMES:
Health-related behaviour | Change from Baseline to end-of-study (6-month)
  Health-related behaviour chosen by the ambassadors (each country could decide to include or not): this outcome will be decided after focus group, considering that SEEDS project is an extreme CS project, and ambassadors should be involved in the whole process and choose at least one of the three outcomes. The tool for evaluating this outcome will be developed for each country after focus groups implementation.
Determinants of each of the behaviours | Change from Baseline to end-of-study (6-month)
  According to the Theory of Planned Behaviour, the main determinants of behaviour are attitude, beliefs, subjective norms and perceived control, which all shape the behavioural intentions. For this purpose, several questions will be included to assess the determinants of behaviours, mainly related to attitudes and environmental factors, also considering the results of the focus groups, according to the guidelines.

OTHER OUTCOMES:
Family information | Change from Baseline to end-of-study (6-month)
  Includes questions from Health Behaviour in School Aged Children (HBSC) validated questionnaire about family, such as: family affluence scale (FAS scale ranges from 0 - low affluence to 9 high affluence), family structure and family meals and, questions about environment like the use of local green space.
Sex | Baseline
  Percentage of males and females
Age | Baseline
  Median age of participants
Grade | Baseline
  Academic course
Level of education | Baseline
  Academic course
Country of birth of the child | Baseline
  Country of birth of the child
Country of birth of the parents | Baseline
  Country of birth of the parents

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Prof., Principal Investigator — University Rovira i Virgili
Locations (4):
- Department of Nutrition & Dietetics, School of Health Science & Education Harokopio University, 70, El Venizelou Ave,, Athens, Kallithea, Greece
- Department of Public Health, Erasmus MC, University Medical Center Rotterdam, P.O. Box, 2040, Rotterdam, The Netherlands, Netherlands
- Institut d'Investigació Sanitaria Pere i Virgili, Reus, Tarragona, Spain
- Children's Health and Exercise Research Centre, Sport and Health Sciences; College of Life and Environmental Sciences, University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Metadata will be published with a DOI (Digital Object Identifier) and data will be made available upon request after signing a data transfer agreement. It may be the case that the requested data could not be shared due to confidentiality obligations. Data will only be available for those that gave consent to use data in projects other than the SEEDS project.
  In the metadata file will be explained what kind of data is in the dataset and how it is possible to get access to the data. This applies for the codified qualitative and quantitative data generated throughout the whole of the SEEDS project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from the project will be under embargo for a period of five years, or it will be immediately made available upon agreement from the SEEDS Consortium. After this period of time, and upon agreement from the Consortium members, the data will be located in a suitable online repository. At the time at which the data is made available through an online repository anyone will be able to access and use it, in keeping with the necessary regulations from the repository.
  Selected curated data in the SEEDS project will be made available to interested third parties or made available on data sharing platforms. Under no circumstances will data that contain any identifying information be offered. All relevant data will be codified.
  There are no restrictions regarding type of analyses
Access Criteria: Once a request is made, responsible members of the Consortium will be contacted to internally discuss each request. Each partner needs to approve the usage of the data collected by their institution before sharing data with other researchers.
  A suitable data repository will be used for the legacy storage of all the relevant data from the SEEDS project. At the time of writing, one is yet to be decided, however, one which has an existing track record of appropriate need provision will be picked.
  All of the data can be viewed using standard issue programs, such as any word processor for the qualitative data, and an appropriate statistical analysis software package for the quantitative data.

REFERENCES:
- [Derived] Queral J, Llaurado E, Wargers A, Jansen W, Manios Y, Senequier A, Williams CA, Vlachopoulos D, Sola R, Tarro L. Comparison of the four co-created interventions to improve snacking and physical activity behaviour in European adolescents: the SEEDS project. BMC Public Health. 2025 Mar 1;25(1):829. doi: 10.1186/s12889-025-22091-x. PMID 40025539
- [Derived] Wargers A, Elphick CM, Molenberg FJM, Senequier A, Manios Y, Mavrogianni C, Murray C, Queral J, Tarro L, Williams CA, Vlachopoulos D, Jansen W. Stakeholder perspectives on the barriers and facilitators of engagement in healthy lifestyle behaviours in underrepresented adolescents: a focus group study from the European SEEDS project. BMC Public Health. 2024 Jul 25;24(1):1988. doi: 10.1186/s12889-024-19419-4. PMID 39054496
- [Derived] Wargers A, Queral J, Molenberg FJ, Tarro L, Elphick CM, Kalogerakou E, Karagiannis A, Llaurado E, Manios Y, Mavrogianni C, Murray C, Vlachopoulos D, Williams CA, Jansen W, Sola R. Citizen Science to improve healthy and active living among adolescents in four European countries: a protocol of the cluster randomised controlled trial of the Science Engagement to Empower aDolescentS (SEEDS) project. BMJ Open. 2023 May 8;13(5):e070169. doi: 10.1136/bmjopen-2022-070169. PMID 37156575